CLINICAL TRIAL: NCT04299399
Title: Corneal Biomechanical Changes and Related Risk Prediction in Allergic Conjunctivitis
Brief Title: Corneal Biomechanical Changes of Allergic Conjunctivitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2019045
Record Dates: First submitted 2020-03-03; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Conjunctivitis, Allergic; Keratoconus
Keywords: Allergic conjunctivitis; Corneal biomechanics; Keratoconus
MeSH Terms: conditions — Conjunctivitis, Allergic; Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- nomal: Corneal biomechanics, corneal topographic parameters, corneal epithelial thickness, tear inflammatory cytokines levels and conjunctival microvascular parameters will be measured, and comparative analysis of biomechanics with other groups will be performed.
- seasonal allergic conjunctivitis(SAC): Eye rubbing frequency, ocular allergy symptom scores, physical sign scores, corneal biomechanics, corneal topographic parameters, corneal epithelial thickness, tear inflammatory cytokines levels and conjunctival microvascular parameters will be measured, and comparative analysis of corneal biomechanics with other groups and correlation analysis of corneal biomechanical parameters and other measurement indicators will be performed.
- vernal keratoconjunctivitis (VKC): At first visit, eye rubbing frequency, ocular allergy symptom scores, physical sign scores, corneal biomechanics, corneal topographic parameters, corneal epithelial thickness, tear inflammatory cytokines levels and conjunctival microvascular parameters will be measured. All patients will adopt a unified medication regimen:0.1% tacrolimus eye drops four times daily; 0.1% flumirone eye drops twice daily; azelastine hydrochloride eye drops four times daily; hyaluronic acid sodium eye drops four times daily. After 1M, 0.1% flumilone eye drops will be replaced with 0.02% flumirone eye drops twice daily, and rest of the medication will remain unchanged. The same ophthalmological examinations will be performed again after 3 month medication.
- keratoconus: Corneal biomechanics, corneal topographic parameters, corneal epithelial thickness, tear inflammatory cytokines levels and conjunctival microvascular parameters will be measured, and comparative analysis of these parameters with other groups will be performed.

SUMMARY:
By measuring and comparing the corneal biomechanical parameters of normal people, patients with allergic conjunctivitis, keratoconus, whether allergic conjunctivitis causes changes in corneal biomechanics can be explored, and sensitive mechanical indicators of allergic conjunctivitis can be identified. Furthermore, through rubbing frequency, ocular allergic symptom scores and physical sign scores observation, corneal morphological parameters, corneal epithelial thickness, tear inflammatory cytokines levels, and conjunctival microvascular parameters measurements, related factors affecting corneal biomechanics in patients with allergic conjunctivitis can be identified. Otherwise, by comparing corneal biomechanical changes in vernal keratoconjunctivitis before and after drug treatment, biomechanical change tendency during treatment can be clarified.

DETAILED DESCRIPTION:
The current study involves 3 parts. The first part aims to explore whether allergic conjunctivitis causes changes in corneal biomechanics and to identify sensitive mechanical indicators of allergic conjunctivitis. This part is a cross-sectional study. Four groups are included: normal group, vernal keratoconjunctivitis (VKC) group, seasonal allergic conjunctivitis (SAC) group and keratoconus (KC) group, with 25 eyes in each group (in normal group one eye is randomly selected , and in VKC group, SAC group and KC group the more severe one is selected). Patients in all groups meet inclusion criteria and voluntarily join this study with informed consents. Medical history is collected, including basic information, allergic history and course of disease. Corneal biomechanics is measured by Corvis ST. The difference of corneal biomechanics among groups is analyzed to determine corneal biomechanical changes of AC and to find sensitive mechanical indicators of AC.

The second part aims to identify related factors affecting corneal biomechanics in patients with allergic conjunctivitis. This part is also a cross-sectional study. Four groups are included: normal group, VKC group, SAC group and KC group, with 25 eyes in each group. Medical history is collected, including basic information, allergic history and course of disease. Eye rubbing frequency, ocular allergic symptom scores and physical sign scores are measured and recorded in VKC group and SAC group. Corneal biomechanics measured by Corvis ST, corneal morphological parameters measured by Pentacam, corneal epithelial thickness measured by Optovue OCT, tear cytokine levels measured by Milliplex kit and conjunctival microvascular parameters measured by functional slit lamp are performed in all patients. Correlation analysis of corneal biomechanical parameters and other measurement indicators in VKC group and SAC group is performed to determine the relevant influencing factors of corneal biomechanics in AC.

The third part aims to determine corneal biomechanical change tendency during treatment in VKC. This part is a prospective case-control study. 25 patients with 25 eyes (the more severe eye is selected) are included. Medical history is collected, including basic information, allergic history and course of disease. Eye rubbing frequency, ocular allergic symptom scores and physical sign scores are measured and recorded in VKC group and SAC group. Corneal biomechanics measured by Corvis ST, corneal morphological parameters measured by Pentacam, corneal epithelial thickness measured by Optovue OCT, tear cytokine levels measured by Milliplex kit and conjunctival microvascular parameters measured by functional slit lamp are performed in all patients before drug treatment. And all the patients adopt a unified medication regimen. The same ophthalmological examinations are performed again after 3 month medication. Based on the analysis of the difference between the two measurements before and after the drug treatment, corneal biomechanical change tendency during treatment in VKC is clarified and the potential mechanical parameter needed to be monitored during follow-up is identified. The specific therapeutic regimen is as follows: 0.1% tacrolimus eye drops four times daily; 0.1% flumirone eye drops twice daily; azelastine hydrochloride eye drops four times daily; hyaluronic acid sodium eye drops four times daily. After 1M, 0.1% flumilone eye drops is replaced with 0.02% flumirone eye drops twice daily, and the rest of the medication remaines unchanged.

ELIGIBILITY:
Normal group

Inclusion Criteria:

1. No abnormalities are found by slit lamp and Pentacam.
2. Diopters: diopter of spherical: -6.0D~+3.0D, diopter of cylinder: -2.0D~+2.0D, spherical equivalent: -6.0D~+3.0D
3. Best corrected visual acuity ≥ 1.0

Exclusion Criteria:

1. Patients diagnosed with other eye diseases other than refractive error.
2. With a history of eye surgery or trauma.
3. With systemic diseases such as immune diseases and connective tissue diseases.
4. With a family history of keratoconus and glaucoma.
5. Wear soft contact lens within 2 weeks or rigid contact lens within 1 month.

SAC group

Inclusion Criteria:

1. Symptoms: Itching, foreign body sensation, increased discharge in conjunctival sac. And children may mainly show an increase in blinking frequency.
2. Signs: conjunctival hyperemia, swelling, tarsal papillae.
3. Medical history: seasonal onset
4. Diopters: diopter of spherical: -6.0D~+3.0D, diopter of cylinder: -2.0D~+2.0D, spherical equivalent: -6.0D~+3.0D
5. Best corrected visual acuity ≥ 0.8

Exclusion Criteria:

1. Corneal scar.
2. Other active inflammatory diseases of the eye.
3. With a history of eye surgery or trauma.
4. With systemic diseases such as immune diseases and connective tissue diseases.
5. Wear soft contact lens within 2 weeks or rigid contact lens within 1 month.
6. Unable to fixate and cooperate.

VKC group

Inclusion Criteria:

1. Symptoms: Itching, foreign body sensation, increased discharge in conjunctival sac. And children may mainly show an increase in blinking frequency.
2. Signs: giant papillae on the upper tarsal conjunctiva and gelatinous infiltration of the limbus.
3. Diopters: diopter of spherical: -6.0D~+3.0D, diopter of cylinder: -2.0D~+2.0D, spherical equivalent: -6.0D~+3.0D
4. Best corrected visual acuity ≥ 0.8

Exclusion Criteria:

The same as SAC group.

Keratoconus group

Inclusion Criteria:

1. With a history of myopia and astigmatism
2. Best corrected visual acuity <1.0
3. At least 1 positive sign of the following is found by slit lamp examination: thinning of the corneal stroma, a cone-shaped ectatic protrusion of the cornea, Fleischer ring and Vogt striae.
4. Typical signs of corneal topography: central corneal power value of the anterior surface >47D, central inferior/superior dioptric asymmetry >3D (within 3mm), central dioptric asymmetry between two eyes >1D.

Exclusion Criteria:

The same as SAC group.

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patients of Zhongshan ophthalmic center and healthy volunteers recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Corneal biomechanics | Baseline in all groups and after 3m medication in VKC group
  The corneal biomechanics parameters are measure by Corvis ST, including A1 Time, A1 Velocity, A2 Time, A2 Velocity, HC Time, PD, DA, SP-A1, CBI, TBI and so on.

SECONDARY OUTCOMES:
Eye rubbing frequency | Baseline in SAC and VKC group, and after 3m medication in VKC group
  According to the frequency of eye rubbing, the scores range from 0 to 5 points, 0 point represents no eye rubbing, 1 point means very few eye rubbing, and 5 points represents eye rubbing all the time.
Ocular allergic symptom scores | Baseline in SAC and VKC group, and after 3m medication in VKC group
  Ocular allergic symptoms are evaluated from six aspects: itching, redness, tearing, foreign body sensation, photophobia, and discharges. The scores range from 0 to 3 according to the severity of each symptom. 0 point means no symptoms, 3 points represents serious symptoms. And the total ocular allergic symptom scores range from 0 to 18.
Ocular sign scores | Baseline in SAC and VKC group, and after 3m medication in VKC group
  Ocular sign scores are evaluated from three major aspects: conjunctiva, limbus and cornea. Conjunctival signs include hyperemia, swelling and tarsal papillae. Limbal signs include swelling and Horner-Trantas dots. Corneal sign is evaluated according to corneal epithelial staining. According to the severity of each sign, the sign scores range from 0 to 3 respectively, with 0 point indicating no corresponding signs and 3 points representing serious signs. And the total ocular sign scores range from 0 to 18.
Morphological parameters of corneal topography | Baseline in all groups and after 3m medication in VKC group
  The morphological parameters are measure by Pentacam, including K1, K2, Km of the front and back surface, astigmatism, ISV, IVA, IHD, KI, CKI, IHA, BAD-D and corneal ocular densitometry.
Corneal epithelial thickness | Baseline in all groups and after 3m medication in VKC group
  The corneal epithelial thickness parameters are measured by RTvue OCT, including corneal thickness map and corneal epithelial thickness map within 9 mm, which are divided into four concentric circles with the diameters of 2mm, 5mm, 7mm and 9mm respectively. And the area between adjacent concentric circles are divided into 8 different areas, including superior, superior-temporal, temporal, temporal-inferior, inferior, inferior-nasal, nasal, and superior-nasal area, with a total of 25 areas.
Conjunctival microvascular parameters | Baseline in all groups and after 3m medication in VKC group
  Conjunctival microvascular parameters are measured by functional slit-lamp biomicroscope，including Va, Vs, Q, Mean Diameter, Dbox and D0.
Tear inflammatory cytokines levels | Baseline in all groups and after 3m medication in VKC group
  Kinds of tear inflammatory cytokines levels are measured, including ITAC, GM-CSF, Fractalkine, IFNy, IL-10, MIP-3a, IL-12(p70), IL-13, IL-17A, IL-1b, IL-2, IL-21, IL-4, IL-23, IL-5, IL-6, IL-7, IL-8, MIP-1a, MIP-1b and TFNa.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yuan, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-Sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Q, Yu F, Feng Z, Li W, Li N, Du X, Zhao X, Li S, Yuan J. Changes in Anterior and Posterior Corneal Elevation in Patients With Allergic Conjunctivitis. Front Med (Lausanne). 2021 Nov 24;8:788302. doi: 10.3389/fmed.2021.788302. eCollection 2021. PMID 34901095
- [Derived] Wang Q, Deng Y, Li S, Du X, Zhao X, Zhang T, Yuan J. Corneal biomechanical changes in allergic conjunctivitis. Eye Vis (Lond). 2021 May 3;8(1):17. doi: 10.1186/s40662-021-00241-7. PMID 33934706